CLINICAL TRIAL: NCT00006103
Title: Interracial Study of CPT-11 (Irinotecan) Pharmacokinetics in 5-Fluorouracil Refractory Colorectal Cancer: A Population Pharmacokinetic/Pharmacodynamic Study of CPT-11
Brief Title: Combination Chemotherapy in Treating Patients With Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9864; U10CA031946 (NIH); CLB-9864; E-C9864; CDR0000068113 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-08-03; First posted 2003-09-03 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Irinotecan; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- irinotecan + leucovorin + fluorouracil (Experimental): Patients receive irinotecan IV over 90 minutes, leucovorin calcium IV, and fluorouracil IV on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for a total of 5 courses in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 3 months for 1 year and then every 6 months thereafter.
  Interventions: Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium

INTERVENTIONS:
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if the effectiveness of irinotecan combined with fluorouracil in treating colorectal cancer varies depending on the patient's racial background.

PURPOSE: Phase III trial to study the effectiveness of irinotecan combined with fluorouracil in treating patients from different racial backgrounds who have colorectal cancer that is advanced, recurrent, metastatic or has not responded to treatment with fluorouracil.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the interracial differences in the pharmacokinetics of irinotecan in combination with fluorouracil in terms of SN-38 glucuronidation and biliary index, and gastrointestinal (GI) toxicity in patients with metastatic, locally advanced, or recurrent colorectal cancer.
* Determine if there is a significant relationship between UGT1A1 genotype (promoter and/or coding region mutation) and CYP3A4 promoter genotype, vs GI toxicity, bone marrow toxicity, and pharmacokinetics of irinotecan in this patient population.

OUTLINE: Patients are stratified according to race (Asian or Pacific Islander vs black vs Hispanic vs white).

Patients receive irinotecan IV over 90 minutes, leucovorin calcium IV, and fluorouracil IV on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for a total of 5 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 400 patients (100 per stratum) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum

  * Metastatic, locally advanced, or recurrent disease
* Patients must have at least 2 generations (parents and grandparents) who belong to one of the following racial groups:

  * Asian or Pacific Islander (e.g., China, Japan, Korea, the Philippine Islands, or Samoa)
  * Black (originating from the black racial groups of Africa)
  * Hispanic (originating from Mexico, Puerto Rico, Cuba, Central or South America, or other Spanish culture)
  * White (originating from the peoples of Europe, North Africa, or the Middle East)
* No patients with parents or grandparents of mixed race or race other than that of the patient

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* CTC 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST no greater than 3 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior adjuvant fluorouracil allowed if relapse occurred at least 6 months after completion of fluorouracil
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No prior irinotecan
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormones except steroids for adrenal failure, hormones for nondisease related conditions (e.g., insulin for diabetes), or intermittent dexamethasone as an antiemetic
* No concurrent prednisone

Radiotherapy:

* At least 4 weeks since prior radiotherapy (except to bone or soft tissue involving less than 25% of bone marrow)
* No concurrent radiotherapy

Surgery:

* At least 4 weeks since prior major surgery

Other:

* No concurrent phenobarbital, valproate, or cyclosporine
* None of the following concurrently during first course of therapy:

  * Macrolide antibiotics (e.g., azithromycin, erythromycin, clarithromycin, troleandomycin, dapsone)
  * Azole antibiotics (e.g., fuconazole, miconazole, itraconazole, ketoconazole)
  * Triazobenzodiazepines (e.g., alprazolam, midazolam, triazolam)
  * Antidepressants (e.g., fluoxetine, setraline hydrochloride, fluoxamine, nefazodone hydrochloride)
  * Quinolone antimicrobials (e.g., ciprofloxacin, ofloxacin)
  * Imidazole antibiotics (e.g., clotrimazole)
  * Anti-ulcer medications (e.g., omeprazole, lansoprazole)
  * Ethinyl estradiol
  * Diltiazem
  * Cimetidine hydrochloride
  * Cisapride
  * Terfenadine
  * Rifampin
  * Glucocorticoids
  * Antiepileptics
  * Grapefruit juice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2000-07; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Brian Leyland-Jones, MD, Study Chair — McGill Cancer Centre at McGill University